CLINICAL TRIAL: NCT00497536
Title: Pharmacokinetics of Insulin Aspart (IAsp) Following Continuous Subcutaneous Insulin Infusion (CSII) in Patients With Type 1 Diabetes Mellitus (T1DM)- Basal Rate Resolution.
Brief Title: Pharmacokinetics of IAsp Following CSII in Patients With T1DM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Charlotte Amalie Ihlo, University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2007-001912-21
Record Dates: First submitted 2007-07-04; First posted 2007-07-06 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus; Continuous Subcutaneous Insulin Infusion (CSII)
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): ≈ bolus protocol.
  Interventions: Drug: Insulin Aspart (IAsp)
- 2 (Active Comparator): ≈ CSII protocol
  Interventions: Drug: Insulin Aspart (IAsp).
- 3 (Active Comparator): ≈ CIII protocol.
  Interventions: Drug: Insulin Aspart (IAsp)

INTERVENTIONS:
Drug: Insulin Aspart (IAsp) — IAsp 100 U.
  ≈ bolus protocol: From 6 pm until 6 am
  • 50 % of habitual 24 hour insulin need/24 hours = basal rate (per hour)
  From 8 am until 6 pm
  1 dose/h + 50 % s.c. (≈ bolus).
  Arms: 1
Drug: Insulin Aspart (IAsp). — IAsp 100 U From 6 pm until 8 am
  • 50 % of habitual 24 hour insulin need/24 hours = basal rate (per hour)
  From 8 am until 6 pm 50 % increase of basal rate
  Arms: 2
Drug: Insulin Aspart (IAsp) — IAsp 100 U From 6 pm until 8 am
  • 50 % of habitual 24 hour insulin need/24 hours = basal rate (per hour)
  From 8 am until 6 pm 50 % increase of basal rate
  Arms: 3

SUMMARY:
The primary objective of the study is to compare SSPIAsp during CSII giving one bolus per hour compared with multiple boluses per hour.

The secondary objective is to compare SSPIAsp during continuous subcutaneous insulin infusion (CSII) versus continuous intravenous insulin infusion (CIII).

DETAILED DESCRIPTION:
Rapid acting insulin, like insulin aspart, can be administered as CSII. The insulin can be administered as a basal rate with additional insulin administration from the pump related to mealtimes.

Insulin is physiologically secreted in a pulsate manner from the pancreatic β-cells with a period of 5-10 minutes, and this is responsible for plasma insulin oscillations with similar frequency. The oscillatory pattern is believed to optimize control mechanisms of insulin to enhance its action on metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (T1DM)
* Insulin pump users' ≥ 48 hours, 24 h dose < 80 U
* Insulin dose ≥ 0,4 IE/kg/24hours
* 18 years < age < 50 years
* Time since diagnosis of T1DM ≥ 5 years
* HbA1c ≤ 8,5 %
* Safe anticonceptive for fertile women
* Being able to understand and read Danish

Exclusion Criteria:

* Dysregulation of endocrine disorders other than type 1 diabetes mellitus
* Severe dysregulation of diabetes mellitus
* Other severe adverse disease
* Pregnancy, planning pregnancy, or nursing

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
CV SSPIasp | 6 hours

SECONDARY OUTCOMES:
• Δ SSPIAsp (S.C. /I.V.) • AUC IAsp • Tmax IAsp • Cmax IAsp - Bioequivalence of Iasp under SS (GIR, S-FFA, S-glycerol) | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Lauritzen, MD, Study Director — University of Aarhus; Torben Laursen, MD, Study Director — University of Aarhus
Locations (1):
- Medicinsk Endokrinologisk Afdeling M, Aarhus C, Central Jutland, Denmark